CLINICAL TRIAL: NCT07281612
Title: A Randomized Controlled Trial Comparing Hand-made Extracorporeal Knotting Versus Clip for Stump Closure in Laparoscopic Appendectomy
Brief Title: Hand-made Extracorporeal Knotting Versus Clip for Stump Closure in Laparoscopic Appendectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Punjab Health Care Commission (Other)
Responsible Party: Principal Investigator, Haseeb Ul Hassan, Doctor, Abbas Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIMS-APP-Knot-vs-Clip
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-03

CONDITIONS: Appendicectomy
Keywords: Appendicectomy; stump closure; knotting; clip; surgery; ileus
MeSH Terms: conditions — Ileus | interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Made Knot Group (Experimental): Appendiceal stump closure using hand-made extracorporeal knotting (modified Tayside knot). Two extracorporeal knots will be applied to secure the appendiceal stump during laparoscopic appendectomy.
  Interventions: Procedure: Hand-made Extracorporeal Knotting
- Arm 2 (Active Comparator): Appendiceal stump closure using a nonabsorbable polymeric Hem-o-lok® clip. One clip is applied at the appendiceal stump and a second clip may be added 2-3 mm above the first if needed
  Interventions: Procedure: Clip Closure

INTERVENTIONS:
Procedure: Hand-made Extracorporeal Knotting — Appendiceal stump closure performed using a hand-made extracorporeal knot (modified Tayside knot technique). Two knots will be applied. Used during laparoscopic appendectomy
  Arms: Hand Made Knot Group
Procedure: Clip Closure — Appendiceal stump closure performed using a nonabsorbable polymeric Hem-o-lok® clip system (Teleflex Medical, USA). The clip is applied to the stump during laparoscopic appendectomy
  Arms: Arm 2

SUMMARY:
Acute appendicitis is one of the most common causes of emergency abdominal surgery. Laparoscopic appendectomy is now widely used because it offers advantages such as shorter hospital stay, less postoperative pain, and better cosmetic outcomes. However, the optimal technique for appendiceal stump closure remains unclear, and different methods such as endoloops, clips, sutures, and staplers are currently used in clinical practice.

This randomized controlled trial will compare two commonly used stump closure techniques during laparoscopic appendectomy: hand-made extracorporeal knotting and polymeric clip application. Participants will be randomly assigned in a 1:1 ratio to either group. The study outcomes include failure of technique, postoperative ileus, and intra-abdominal infection within 15 days after surgery.

The aim of this study is to determine whether hand-made extracorporeal knotting is more effective than clip application in reducing postoperative complications related to appendiceal stump closure.

DETAILED DESCRIPTION:
Acute appendicitis is a major cause of acute abdomen and a frequent indication for emergency surgery. Laparoscopic appendectomy has become the preferred surgical approach due to advantages such as reduced postoperative pain, quicker recovery, lower wound infection rates, and improved cosmetic outcomes. Despite technical advancements, appendiceal stump leakage remains a serious postoperative concern, potentially resulting in intra-abdominal sepsis and reoperation.

A variety of appendiceal stump closure techniques are in use, including endoloops, sutures, staplers, and clips. Both hand-made extracorporeal knotting and polymeric nonabsorbable clips (Hem-o-lok®) are commonly employed and considered safe. Hand-made extracorporeal knotting has potential advantages of lower cost and usability in resource-limited settings, but the optimal closure technique remains controversial and evidence is limited.

This study is designed as a single-center, prospective, parallel-group randomized controlled trial conducted at Abbas Institute of Medical Sciences, Muzaffarabad. A total of 190 patients aged 10-70 years presenting with acute appendicitis and undergoing laparoscopic appendectomy will be enrolled. After diagnostic laparoscopy and confirmation of eligibility, participants will be randomized by simple lottery method into one of two groups:

Intervention Group: appendiceal stump closure using hand-made extracorporeal knotting (modified Tayside knot), with two knots applied.

Comparator Group: appendiceal stump closure using a nonabsorbable polymeric Hem-o-lok® clip.

Demographic variables, comorbidities, stump diameter, and operative time will be recorded. Outcomes will be assessed intraoperatively and postoperatively, with follow-up continuing until postoperative day 15. The primary outcome is intra-abdominal infection within 15 days. Secondary outcomes include failure of technique during surgery and postoperative ileus.

Statistical analysis will be performed using SPSS software. Categorical variables will be analyzed using a chi-square test, and continuous variables will be summarized as mean ± standard deviation. A p-value ≤ 0.05 will be considered statistically significant.

The findings of this trial may help determine whether hand-made extracorporeal knotting provides superior clinical outcomes or cost advantages compared to polymeric clips, and may guide standardization of appendiceal stump closure techniques in laparoscopic appendectomy, particularly in low-resource surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 to 70 years
* Either sex
* Clinical diagnosis of acute appendicitis with Alvarado score >6
* ASA physical status I-III
* Planned laparoscopic appendectomy

Exclusion Criteria:

* Patient request for open appendectomy
* Complicated appendicitis (perforation, appendicular abscess, or appendicular mass)
* Local or diffuse peritonitis
* Friable or necrotic appendix base
* Pelvic inflammatory disease

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Post operative ileus | within 48 hours of surgery
  Postoperative ileus defined as absence of bowel movement, passage of flatus, or audible bowel sounds up to 48 hours after surgery
Intra abdominal infection | within 15 days of surgery
  Intra-abdominal infection defined as presence of fever, abdominal pain, or systemic symptoms confirmed by CT scan showing intra-abdominal abscess or infection requiring medical or surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Haseeb Ul Hassan, MBBS, Principal Investigator — AIMS Institute
Locations (1):
- AIMS, Muzaffarabad, AJK/Punjab, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
At this time, plans for sharing individual participant data (IPD) have not been finalized. Data access may be limited due to patient privacy considerations, lack of a secure data-sharing framework, and institutional policies regarding confidentiality. If future sharing becomes possible, a detailed plan will be provided.